CLINICAL TRIAL: NCT01162161
Title: Role of Sphingolipids in Pulmonary Edema
Acronym: 09-045
Status: Completed | Type: Observational
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Other Study IDs: Sphingo-AC
Record Dates: First submitted 2010-07-13; First posted 2010-07-14 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Pulmonary Edema
Keywords: sphingolipid; ceramide; sphingomyelinase
MeSH Terms: conditions — Pulmonary Edema

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- hydrostatic pulmonary edema: patients with a pulmonary edema caused by chronic heart failure
- toxic pulmonary edema: patients with a pulmonary edema preceded by pneumonia
- control group: not ventilated patients without any pulmonary edema receiving a bronchoscopy due to another pulmonary problem (no pneumonia, no heart failure)

SUMMARY:
In this mono-center prospective study, the impact of changes in the sphingolipid metabolism in patients with pulmonary edema will be investigated.

DETAILED DESCRIPTION:
There will be three groups of patients:

1. hydrostatic pulmonary edema
2. toxic pulmonary edema
3. not ventilated patients without any pulmonary edema

Samples of a routine bronchoalveolar lavage and EDTA-blood will be analysed in respect of sphingolipids, ceramide, sphingomyelin-phosphodiesterase and several cytokines.

ELIGIBILITY:
Inclusion Criteria:

* above the age of 18

Exclusion Criteria:

* taking steroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 3 groups
  first group: patients with a lung oedema because of a pneumonia (about 30 patients)
  second group: patients with a lung oedema because of cardiac insufficiency (about 25 patients)
  third group: patients without any lung oedema (about 15 patients)
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2010-07; Primary Completion 2012-12 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Krüger, MD, PhD, Principal Investigator — RWTH Aachen University
Locations (1):
- Medical Clinic I, University Hospital Aachen, Aachen, North Rhine-Westphalia, Germany